CLINICAL TRIAL: NCT05295017
Title: LEVANTIS-0093A: GAGomes for Multi-Cancer Early Detection in High-Risk Adults (LEV93A)
Acronym: LEV93A
Status: Active, not recruiting | Type: Observational
Sponsor: Elypta (Industry)
Responsible Party: Sponsor
Other Study IDs: GR 22-016
Record Dates: First submitted 2022-02-14; First posted 2022-03-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cancer
Keywords: liquid biopsy; multi-cancer early detection; glycosaminoglycans
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Prospectively collected blood samples sourced from patients enrolled in study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
LEVANTIS-0093A (LEV93A) is a prospective cohort observational clinical study to validate the plasma free GAGome MCED test in adults at high risk of developing cancer ("high-risk adults"), specifically in 55-80-year-old adults with significant smoking history.

LEV93A will use plasma biospecimens collected within the Yorkshire Lung Screening Trial Biomarker sub-study and corresponding participant data prospectively collected within the Yorkshire Lung Screening Trial (YLST) and the Yorkshire Kidney Screening Trial (YKST) all of which are sponsored by the University of Leeds and funded by Yorkshire Cancer Research (Award references: L403, L403B L403C), in collaboration with the University of Leeds, with the University of Manchester and with the Leeds Teaching Hospitals.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 55-80 years old
* Significant smoking history, defined as current or ex-smokers and any of the following criteria:

  * 30 pack year history of smoking and current smoker or quit within the last 15 years (USPSTF criteria).
  * Lung cancer risk of ≥1.51% over 6 years as calculated by the PLCOM2012 score
  * Lung cancer risk of ≥5% over 5 years as calculated by the LLPv2. Score
* Consenting to participate to both YLST and YLST Biomarker trials
* Able to donate a blood sample

Exclusion Criteria

* Deemed medically unfit for sample collection
* Contraindication for study procedures or sampling
* Not consenting to participate to YKST trial

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults between 55 and 80 years old with significant smoking history ("high-risk adults").
Sampling Method: Probability Sample
Enrollment: 1235 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the plasma free GAGome MCED test | Within 365 days after the biosampling visit
  Indicative of any-type cancer vs. no cancer diagnosis

SECONDARY OUTCOMES:
Accuracy to the "putative cancer location" (PCL) model among cases (confirmed cancer diagnosis) | Within 365 days after the biosampling visit
  Accuracy to the "putative cancer location" (PCL) model among cases (confirmed cancer diagnosis)
Sensitivity and specificity of the plasma free GAGome MCED test followed by low-dose computed tomography (LDCT) | Within 365 days after the biosampling visit
  Indicative of any-type cancer vs. no cancer diagnosis in combination with LDCT
Sensitivity and specificity of LDCT followed by plasma free GAGome MCED test | Within 365 days after the biosampling visit
  Indicative of any-type cancer vs. no cancer diagnosis in combination with LDCT

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Gatto, PhD, Principal Investigator — Elypta AB
Locations (1):
- Leads Teaching Hospitals Trust, Leeds, United Kingdom